CLINICAL TRIAL: NCT06152666
Title: Understanding Enablers, Barriers, and Unexpected Outcomes Associated With Adoption of Routine Day-case Surgery Pathways for Common Endourology Operations: Qualitative Interviews With Healthcare Professionals.
Brief Title: Day-case Endourology; Enablers, Barriers, Unexpected Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: Royal Cornwall Hospitals Trust (Other); North Bristol NHS Trust (Other); Gloucestershire Hospitals NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other); Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 326803
Record Dates: First submitted 2023-11-21; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Bladder Cancer; Bladder Outlet Obstruction; Urolithiasis
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urinary Bladder Neck Obstruction; Urolithiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Staff: Members of healthcare teams involved in the delivery of day-case endourology operations.
  Interventions: Other: None - qualitative interviews

INTERVENTIONS:
Other: None - qualitative interviews — These are qualitative interviews and involve no intervention

SUMMARY:
A qualitative research study conducted in hospitals across England, in which staff members will be interviewed. We will interview staff who are directly or indirectly involved in delivering care for patients undergoing the operations of interest; namely bladder tumour resection, prostate resection or enucleation, and ureteroscopy for upper urinary tract stones. We hope to find out the reasons why some hospitals can perform day-case surgery with very high rates, and why others do not. We also hope to find out about any unexpected outcomes observed when performing day-case surgery for the operations of interest.

Staff working in a range of different hospitals from across England with varying day-case rates will be interviewed. Hospitals in large city and more rural areas will be assessed. Interviews are anticipated to take place over a six month period. The study will end when "saturation" is achieved, whereby no new themes are identified through interviews. Saturation will be sought for each individual operation of interest.

DETAILED DESCRIPTION:
Safe day-case surgery pathways offer to reduce pressure on hospitals by avoiding overnight inpatient admission. This is particularly relevant given the intense pressures on hospital resources in the United Kingdom. Urological surgery includes a number of frequently performed operations for which safe day-case surgery pathways have been demonstrated. These include bladder tumour resection (TURBT), prostate resection or enucleation using diathermy or laser (TURP and TUEP), and ureteroscopy and laser for upper urinary tract stones (URS). All of these operation types involve endoscopic access to the bladder via the urethra, and do not involve skin incisions. They can be performed under general or spinal anaesthesia, although spinal anaesthesia is rarely used for ureteroscopy.

For the 12 months from December 2021, the national median day-case rate for transurethral resection of bladder tumour In England was 21.1%, and ranged from 0% to 87.3% at different hospitals, with an interquartile range (IQR) of 10.5% to 37.7%, and 23,071 cases performed in total. For bladder outflow obstruction surgery the median day-case rate was 7.7% (range 0% to 82.4%, IQR 4.4% to 19.1%, 18,912 cases), and this includes TURP and TUEP. For URS the median day case rate was 60.1% (range 0% to 87.9%, IQR 44.4% to 69.7%, 23,130 cases). This demonstrates that for these common operations there is significant variation in practice across England.

The Getting It Right First Time (GIRFT) Urology programme advocates for a "day-case by default" approach to TURBT and URS, and that day-case surgery should ideally be offered for prostate resection and enucleation. As well as reducing pressure on inpatient services, greater day-case adoption offers to reduce financial costs, shorten waiting lists by allowing greater access to day-case theatres away from the acute hospital, and reduce environmental impact by adopting a less resource-intensive approach. It also offers a more standardised patient experience.

National day-case rates for all of TURBT, TURP/TUEP and URS have increased over the past five years, however the wide variation in practice identifies a need to understand reasons underlying a significant observed divergence in practice. We want to understand why some hospitals have rapidly adopted day-case surgery whereas others have not. Furthermore, it is necessary to understand any positive and negative outcomes associated with the increased utilisation of day-case surgery. In order to explore this area we intend to perform qualitative research involving members of staff involved in the delivery of one or more of the operations of interest. We will interview staff from a range of different hospitals with differing day-case performances to further understand enablers and barriers associated with day-case adoption. We would also like to understand staff members' experiences of any wider unexpected outcomes associated with day-case surgery adoption.

ELIGIBILITY:
Inclusion Criteria:

* Staff members who are routinely involved, either directly or indirectly, in the delivery of any of TURBT, TURP, TUEP, URS within NHS hospitals.
* Willing and able to provide informed consent

Exclusion Criteria:

* Staff who are not regularly involved in any of TURBT, TURP, TUEP or URS, defined as being involved in the operation less than 10 cases per year.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Any of the following staff members from across a range of urology units:
  * Consultant and trainee urologists
  * Anaesthetists
  * Theatre nursing staff and healthcare assistants
  * Day-case unit nursing staff
  * Inpatient ward nursing staff
  * Cancer nurse specialists
  * Urology managers
  * Urology department clinical leads
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Staff perspectives on delivering day-case endourology surgery | 6 months
  Obtained through qualitative interview

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Devon University Healthcare NHS Foundation Trust, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
None. Anonymised quotes will be used in the published study report.

DOCUMENTS (1):
  • Study Protocol (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT06152666/Prot_000.pdf